CLINICAL TRIAL: NCT06122727
Title: Comparison of Customized and Standard Total Knee Replacements: a Pilot Study
Brief Title: Comparison of Custom and Standard Total Knee Replacements
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3POD-TKA
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CUSTOM (Experimental): patients will undergo primary TKA by implanting a prosthetic model (YourKnee, Rejoint) with a design specifically based on each patient's real knee morphology and using PSI surgical technique and instrumentation.
  Interventions: Procedure: total knee arthroplasty
- TRADITIONAL (Active Comparator): patients will undergo a primary TKR by implanting a prosthetic model of the same standard design for all using the usual surgical technique and instrumentation (based on the use of the guided intramedullary femur and extramedullary tibia).
  Interventions: Procedure: total knee arthroplasty

INTERVENTIONS:
Procedure: total knee arthroplasty — In detail, in the STANDARD group, patients will undergo a primary TKR by implanting a prosthetic model of the same standard design for all using the usual surgical technique and instrumentation (based on the use of guide intramedullary of femur and extramedullary of tibia); in the PERSONALIZED group, patients will undergo a primary TKA by implanting a prosthetic model (YourKnee, Rejoint) with design based specifically on each patient's actual knee morphology and using PSI surgical technique and instrumentation. In both groups, the approach of the basic prosthetic design base will be of the Cruciate-Retaining (CR) type with congruent polyethylene (PE), with standard and customized for the STANDARD and CUSTOM group, respectively.

SUMMARY:
Total knee arthroplasty (TKA) is the most common surgery in North America and the second most common in Europe. One of the most critical issues for stability and durability of the interventional is the prosthesis-bone geometric fit, where a required a perfect match; the recent availability of custom 3D implants can overcome this problem. In order to further improve a TKA surgery, it is in fact, it is possible today to completely customize the procedure for each individual patient, with cost and time now accessible. This intervention can be performed with the use of instrumentation specific to the patient (so-called resin 'cutting templates' referred to as PSI, "Patient Specific Instrumentation") to make cuts accurate bone cuts in accordance with a specific 3D preoperative plan . Also the design and fabrication in of the components prosthetic components themselves, in metal and polyethylene, is done by means of 3D printing. Based on the unique anatomy of each patient, the precise sagittal orientation and axial rotation of the components of the prosthesis customized for the surgeon, it is possible to plan and perform the surgery quickly and in accordance with the exact specifications of the individual patient. These procedures should also make it possible to greatly reduce the instrumentation and the sizes that need to be available in the operating room, reducing time and costs associated with transportation and storage . The objective of this study is to compare primary TKAs performed with a customized procedure (prostheses customized for each patient based on his or her reconstructed knee morphology by tomographic scans, and implanted via cutting guides customized for the patient) with standard primary TKAs, considering: the objective radiological results, the subjective results of the patients and the costs of both procedures.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects older than 40 years and younger than 70 years (≥ 40 age ≤ 70 years) candidates for primary cemented total knee replacement.
* Consenting patients and able to complete scheduled study procedures and follow-up evaluations.
* Patients who have signed the "informed consent" approved by the Ethics Committee.

Exclusion Criteria:

* Social conditions (homeless patients, with restrictions on personal freedom)
* ASA 3
* Deep venous insufficiency Lower limbs
* History of Erisipelas lower limbs
* Neurological or psychocognitive disorders
* Neurological diseases
* Post-traumatic arthritis
* Axial deformities of the knee >10°
* Personal or family history of DVT or EP
* Prosthetic and/or arthrodesis surgeries at another joint of the lower extremities lower limb except that candidate for knee prosthesis
* Pregnant women
* Patients with rheumatic diseases

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Angle Hip Knee Ankle | at baseline (day 0)
  Evaluate by how many degrees the angle HKA (angle obtained by joining the center of rotation of the knee with that of the hip and ankle) planned (desired value) differs from that measured postoperatively (obtained value) When implanting a customized primary TKA (PERSONALIZED group) vs. a standard primary TKA (STANDARD group) according to normal surgical practice.
Angle Hip Knee Ankle | 12 months
  Evaluate by how many degrees the angle HKA (angle obtained by joining the center of rotation of the knee with that of the hip and ankle) planned (desired value) differs from that measured postoperatively (obtained value) When implanting a customized primary TKA (PERSONALIZED group) vs. a standard primary TKA (STANDARD group) according to normal surgical practice.

SECONDARY OUTCOMES:
Visual analogic scale | at baseline (day 0)
  The VAS scale is an objective method of pain measurement
Visual analogic scale | after 3 months
  The VAS scale is an objective method of pain measurement
Visual analogic scale | after 6 months
  The VAS scale is an objective method of pain measurement
Visual analogic scale | after 12 months
  The VAS scale is an objective method of pain measurement
Visual analogic scale | after 24 months
  The VAS scale is an objective method of pain measurement
New Knee Society Score | at baseline (Day 0)
  The KSS contains questions in 2 sections: knee joint (pain, range of motion, stability) and function (walking distance, ability to climb stairs). When calculating the score, deductions are taken for assistive devices and flexion contractures, misalignment, or extension lag.
New Knee Society Score | after 3 months
  The KSS contains questions in 2 sections: knee joint (pain, range of motion, stability) and function (walking distance, ability to climb stairs). When calculating the score, deductions are taken for assistive devices and flexion contractures, misalignment, or extension lag.
New Knee Society Score | after 6 months
  The KSS contains questions in 2 sections: knee joint (pain, range of motion, stability) and function (walking distance, ability to climb stairs). When calculating the score, deductions are taken for assistive devices and flexion contractures, misalignment, or extension lag.
New Knee Society Score | after 12 months
  The KSS contains questions in 2 sections: knee joint (pain, range of motion, stability) and function (walking distance, ability to climb stairs). When calculating the score, deductions are taken for assistive devices and flexion contractures, misalignment, or extension lag.
New Knee Society Score | after 24 months
  The KSS contains questions in 2 sections: knee joint (pain, range of motion, stability) and function (walking distance, ability to climb stairs). When calculating the score, deductions are taken for assistive devices and flexion contractures, misalignment, or extension lag.
Knee injury & Osteoarthritis Outcome Score | at baseline (Day 0)
  The KOOS is self-administered and assesses five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life
Knee injury & Osteoarthritis Outcome Score | after 3 months
  The KOOS is self-administered and assesses five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life
Knee injury & Osteoarthritis Outcome Score | after 6 months
  The KOOS is self-administered and assesses five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life
Knee injury & Osteoarthritis Outcome Score | after 12 months
  The KOOS is self-administered and assesses five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life
Knee injury & Osteoarthritis Outcome Score | after 24 months
  The KOOS is self-administered and assesses five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life
Forgotten Joint Score | at baseline (day 0)
  a patient-reported outcome measure intended to determine a patient's ability to "forget" about their affected joint after surgery or treatment
Forgotten Joint Score | after 3 months
  a patient-reported outcome measure intended to determine a patient's ability to "forget" about their affected joint after surgery or treatment
Forgotten Joint Score | after 6 months
  a patient-reported outcome measure intended to determine a patient's ability to "forget" about their affected joint after surgery or treatment
Forgotten Joint Score | after 12 months
  a patient-reported outcome measure intended to determine a patient's ability to "forget" about their affected joint after surgery or treatment
Forgotten Joint Score | after 24 months
  a patient-reported outcome measure intended to determine a patient's ability to "forget" about their affected joint after surgery or treatment

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Lubbeke A, Silman AJ, Barea C, Prieto-Alhambra D, Carr AJ. Mapping existing hip and knee replacement registries in Europe. Health Policy. 2018 May;122(5):548-557. doi: 10.1016/j.healthpol.2018.03.010. Epub 2018 Mar 17. PMID 29598886
- [Result] Qiu B, Liu F, Tang B, Deng B, Liu F, Zhu W, Zhen D, Xue M, Zhang M. Clinical Study of 3D Imaging and 3D Printing Technique for Patient-Specific Instrumentation in Total Knee Arthroplasty. J Knee Surg. 2017 Oct;30(8):822-828. doi: 10.1055/s-0036-1597980. Epub 2017 Jan 25. PMID 28122388
- [Result] Brinkmann EJ, Fitz W. Custom total knee: understanding the indication and process. Arch Orthop Trauma Surg. 2021 Dec;141(12):2205-2216. doi: 10.1007/s00402-021-04172-9. Epub 2021 Oct 15. PMID 34652517
- [Result] Scuderi GR, Bourne RB, Noble PC, Benjamin JB, Lonner JH, Scott WN. The new Knee Society Knee Scoring System. Clin Orthop Relat Res. 2012 Jan;470(1):3-19. doi: 10.1007/s11999-011-2135-0. No abstract available. PMID 22045067